CLINICAL TRIAL: NCT01597414
Title: Pertuzumab + Trastuzumab (PH) Versus PH Plus Metronomic Chemotherapy (PHM) in the Elderly HER2+ Metastatic Breast Cancer Population Who May Continue on T-DM1 Alone Following Disease Progression While on PH / PHM: an Open-label Multicentre Randomized Phase II Selection Trial of the EORTC Elderly Task Force and Breast Cancer Group
Brief Title: Elderly Metastatic Breast Cancer: Pertuzumab-Herceptin vs Pertuzumab-Herceptin-Metronomic Chemotherapy, Followed by T-DM1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-75111-10114; 2011-006342-32 (EudraCT Number)
Record Dates: First submitted 2012-05-07; First posted 2012-05-14 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Elderly Metastatic Breast Cancer Population
MeSH Terms: interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pertuzumab + trastuzumab (PH) (Active Comparator): Pertuzumab + trastuzumab. After progression,patients will be given the option of receiving T-DM1
  Interventions: Drug: Pertuzumab + trastuzumab
- PH + metronomic chemotherapy (PHM) (Experimental): Pertuzumab + trastuzumab + metronomic chemotherapy. After progression,patients will be given the option of receiving T-DM1
  Interventions: Drug: Pertuzumab + trastuzumab + metronomic chemotherapy

INTERVENTIONS:
Drug: Pertuzumab + trastuzumab — Trastuzumab: loading dose of 8 mg/kg of body weight on cycle 1, followed by a maintenance dose of 6 mg/kg every 3 weeks.
  Pertuzumab: loading dose of 840 mg on cycle 1, followed by 420 mg for subsequent cycles, every 3 weeks.
  if T-DM1: 3.6 mg/kg IV, every 3 weeks.
  Arms: Pertuzumab + trastuzumab (PH)
Drug: Pertuzumab + trastuzumab + metronomic chemotherapy — Pertuzumab and trastuzumab will be administered as in arm A. Cyclophosphamide: daily dose of 50 mg/day. if T-DM1: as in arm A
  Arms: PH + metronomic chemotherapy (PHM)

SUMMARY:
Chemotherapy and HER2 targeted agents can improve survival significantly in metastatic breast cancer. Chemotherapy however is associated with significant side-effects and can impact on Quality of Life and functionality in older patients.

The investigators aim to establish HER2 targeted regimens with minimal toxicity in order to delay or even avoid the use of classical chemotherapy because of competing risks of death in this frail/elderly patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven HER-2 positive
* Newly diagnosed or recurrent (after surgery) stage IV disease (TNM/AJCC v.7).
* Patients must have measurable (RECIST v. 1.1) or evaluable disease
* Performance status (PS) 0-3 (WHO)
* Age ≥ 70 years of age, or ≥ 60 years old with required number of dependencies
* Life expectancy of more than 12 weeks
* Previous adjuvant chemotherapy/anti HER-2 therapy after surgery is allowed, given that the time interval from end of previous treatment to initiation of treatment for metastatic disease is ≥ 6 months.
* Up to one line of anti-HER therapy (trastuzumab or lapatinib) is allowed in combination with hormone therapy for hormone sensitive metastatic breast cancer.
* Adequate organ function
* Before patient randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* No brain metastases that are untreated, symptomatic, or require steroids to control symptoms; or any radiation, surgery, or other therapy to control symptoms from brain metastases within 2 months prior to the first study treatment.
* No prior chemotherapy for metastatic disease is allowed
* No prior treatment with pertuzumab is allowed
* No history of exposure to the following cumulative doses of anthracyclines:
* Doxorubicin or liposomal doxorubicin > 360 mg/m2
* Epirubicin > 720 mg/m2
* Mitoxantrone > 120 mg/m2
* Idarubicin > 90 mg/m2
* If another anthracycline or more than 1 anthracycline has been used, then the cumulative dose must not exceed the equivalent of 360 mg/m2 of doxorubicin.
* No history of palliative radiotherapy within 14 days of randomization
* No history of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or basal cell or spinocellular carcinoma of the skin
* No current uncontrolled hypertension (persistent systolic > 180 mmHg and/or diastolic > 100 mmHg)
* No LVEF below 50%
* No history of significant cardiac disease defined as:
* Symptomatic CHF (NYHA classes II-IV)
* High-risk uncontrolled arrhythmias
* History of myocardial infarction within 6 months prior to randomization
* Clinically significant valvular heart disease
* No angina pectoris requiring anti-angina treatment
* No peripheral neuropathy of Grade ≥ 3 per NCI CTCAE version 4.0.
* No current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures, known infection with HIV, active hepatitis B and/or hepatitis C virus)
* No major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* No history of receiving any investigational treatment within 28 days of randomization
* No history of intolerance (including Grade 3-4 infusion reaction) to trastuzumab
* No unwillingness or inability to comply with the requirements of the protocol as assessed by the investigator
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-03 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate | 6 months after patients in

SECONDARY OUTCOMES:
Overall survival
Breast cancer specific survival
Tumor response rate as measured by RECIST v1.1
Evolution of HRQoL as assessed by EORTC QLQ-C30 and ELD 14 | Up to 1 year after treatment start
Evolution of geriatric assessment | Up to 1 year after treatment start
if T-DM1: progression free survival rate | 6 months after start of T-DM1 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hans Wildiers, MD, Study Chair — UZ Leuven, Leuven, Belgium
Locations (30):
- Belgium (10):
  - UZ Antwerpen, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - Hopital De Jolimont, Haine-Saint-Paul
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven
  - CHU Sart-Tilman, Liège
  - Clinique et Maternité Sainte Elisabeth, Namur
  - AZ Damiaan, Ostend
  - AZ Nikolaas, Sint-Niklaas
- France (4):
  - Centre Georges-Francois-Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Hopital Rene Huguenin - Institut Curie, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
- Italy (2):
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Oncologico Veneto IRCCS - Ospedale Busonera, Padua
- Netherlands (2):
  - Leiden University Medical Centre, Leiden
  - VieCuri - Medisch Centrum voor Noord-Limburg - Locatie Venlo, Venlo
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- Portugal (2):
  - Champalimaud Cancer Center, Lisbon
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon
- Sweden (4):
  - Sahlgrenska Universitetssjukhuet, Gothenburg
  - Ryhov County Hospital, Jönköping
  - Uppsala University Hospital - Akademiska Sjukhuset, Uppsala
  - Vastmanland Centralsjukhuset Vasteras, Västerås
- United Kingdom (5):
  - Velindre NHS Trust - Velindre Cancer Centre, Cardiff
  - NHS Lothian - Western General Hospital, Edinburgh
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Peterborough and Stamford Hospitals NHS Foundation Trust - Peterborough City Hospita, Peterboroug
  - University Hospital Southampton NHS Foundation Trust - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Wildiers H, Tryfonidis K, Dal Lago L, Vuylsteke P, Curigliano G, Waters S, Brouwers B, Altintas S, Touati N, Cardoso F, Brain E. Pertuzumab and trastuzumab with or without metronomic chemotherapy for older patients with HER2-positive metastatic breast cancer (EORTC 75111-10114): an open-label, randomised, phase 2 trial from the Elderly Task Force/Breast Cancer Group. Lancet Oncol. 2018 Mar;19(3):323-336. doi: 10.1016/S1470-2045(18)30083-4. Epub 2018 Feb 9. PMID 29433963